CLINICAL TRIAL: NCT05236816
Title: Relationship Between Hip Abductor Strength and Ankle Stability
Acronym: HIAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021/655
Record Dates: First submitted 2021-12-17; First posted 2022-02-11 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Fatigue
Keywords: Balance; Ankle; Destabilization; Prevention; Hip fatigue
MeSH Terms: conditions — Fatigue | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy (Experimental): Subjects were evaluated before and after a fatiguing exercise of hip abductor muscles that consisted to repeat hip abduction with rate and range of motion until a target decrease of force is attempt
  Interventions: Other: Fatigue (physical exercise)

INTERVENTIONS:
Other: Fatigue (physical exercise) — Subjects were evaluated before and after a fatiguing exercise of hip abductor muscles that consisted to repeat hip abduction with rate and range of motion until a target decrease of force is attempt

SUMMARY:
Ankle sprains are one of the most common injuries in sports. The analysis of risk factors is a priority in order to guide rehabilitation and prevention programs. Among risk factors identified in the literature, weakness of the hip abductor muscles represent a factor favoring recurrent ankle sprains. However, only few studies have investigate the link between the strength of the hip abductor muscles and the deficits in stabilization of the ankle joint. Furthermore, these few studies analysed landing task or undisturbed balance task. It would be interesting to further understand the impact and role of hip abductor muscles on ankle stability during specific ankle-destabilizing task.

The main objective of this study is to establish a link between the strength of the hip abductor muscles and the dynamic postural control performance measured by the modified Star Excursion Balance Test (SEBTm). Secondly, it will be necessary to study the kinematic and neuromuscular control characteristics of the ankle during 4 functional tests:

* SEBTm
* Static unipodal balance
* Weight-bearing inversion test
* Weight-bearing eversion test

These tests will be realized with an ankle destabilizing device. The device is a sandal equipped of an articulator under the rear foot which allow movements in inversion and eversion. Furthermore, tests are realized two times, before and immediatly after a fatiguing exercise. The fatiguing exercise consists to implemented local fatigue on hip abductor muscles by repeating abductions.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18 and 35 years old
* Subject's non-opposition to participate in the study
* Practicing regular physical activity (> 2 hours per week)
* No contraindication to carrying out the protocol
* Affiliation to a French social security scheme or beneficiary of such a scheme

Exclusion Criteria:

* Males or females under 18 or over 35 years
* History of lower limb injuries in the 6 months preceding the protocol
* Diagnosis of chronic ankle instability
* Subject unlikely to cooperate with the study and / or weak cooperation anticipated by the investigator
* Subject's opposition to participating in the study
* Subject without health insurance
* Pregnant woman

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
Surface Electromyography intensity change | 5 minutes before physical exercise
  Measure of muscles activity if peroneus longus and brevis, tibialis anterior, gluteus medius and gastrocnemuis lateralis using wireless and surface electrodes fixed with strap on the skin of subjects
Surface Electromyography intensity change | 5 minutes after physical exercise
  Measure of muscles activity if peroneus longus and brevis, tibialis anterior, gluteus medius and gastrocnemuis lateralis using wireless and surface electrodes fixed with strap on the skin of subjects
Frontal inclination of ankle change | 5 minutes before physical exercise
  Measure of accelerations of ankle joint during tests using inertial measurement unit
Frontal inclination of ankle change | 5 minutes after physical exercise
  Measure of accelerations of ankle joint during tests using inertial measurement unit
SEBT performances change | 5 minutes before physical exercise
  Performances (distance in cm) attempted in each direction of the dynamic postural test
SEBT performances change | 5 minutes after physical exercise
  Performances (distance in cm) attempted in each direction of the dynamic postural test
Hip abductor strength change | 5 minutes before physical exercise
  Measure of maximal isometric strength with a S-shape force transducer
Hip abductor strength change | 5 minutes after physical exercise
  Measure of maximal isometric strength with a S-shape force transducer
Angular velocity of ankle change | 5 minutes before physical exercise
  Measure of angular velocity of ankle joint during tests using inertial measurement unit
Angular velocity of ankle change | 5 minutes after physical exercise
  Measure of angular velocity of ankle joint during tests using inertial measurement unit

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon, Besançon, France

REFERENCES:
- [Result] Dury J, Ravier G, Michel F. Hip Abductor Muscle Fatigue Induces Different Strategies During Disrupted Postural Control. Front Sports Act Living. 2022 Jun 29;4:918402. doi: 10.3389/fspor.2022.918402. eCollection 2022. PMID 35847456
- See also: Hip Abductor Muscle Fatigue Induces Different Strategies During Disrupted Postural Control — https://www.frontiersin.org/journals/sports-and-active-living/articles/10.3389/fspor.2022.918402/full